CLINICAL TRIAL: NCT04190966
Title: A Trial to Study the Effectiveness of Smoking Cessation in the Surgical Pathway Before Major Lung Surgery: Project MURRAY Feasibility Study
Brief Title: Smoking Cessation in the Surgical Pathway Before Major Lung Surgery
Acronym: MURRAY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Birmingham (Other)
Collaborators: University College, London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Worktribe 843842
Record Dates: First submitted 2019-11-28; First posted 2019-12-09 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Smoking Cessation; Thoracic Surgery
Keywords: Postoperative Pulmonary Complications; Smoking Cessation Intervention
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrated smoking cessation (Active Comparator): Integrated smoking cessation delivered by trained health-care practitioners in the thoracic surgical pathway: a three part package of behaviour interventions and pharmacotherapy as per NICE/NCSCT guidance which is supported by an adjunct web-based application.
  Interventions: Behavioral: Integrated Behavioural therapy; Drug: Integrated Pharmacotherapy; Device: Integrated Web-based application
- Usual care smoking cessation (No Intervention): Usual care of standard community/hospital based NHS smoking cessation.

INTERVENTIONS:
Behavioral: Integrated Behavioural therapy — Integrated smoking cessation behavioural therapy
  Arms: Integrated smoking cessation
Drug: Integrated Pharmacotherapy — Integrated smoking cessation pharmacotherapy including choice of combination nicotine replacement therapy, varenicline or electronic cigarettes
  Arms: Integrated smoking cessation
Device: Integrated Web-based application — Integrated smoking cessation web-based application
  Arms: Integrated smoking cessation

SUMMARY:
This is a feasibility study of a personalised, integrated smoking cessation in the surgical pathway in patients undergoing major elective thoracic surgery when compared to usual care of standard community/hospital based NHS smoking cessation. Half the patients will receive the intervention and half the patients will receive usual care.

DETAILED DESCRIPTION:
Smoking prior to major thoracic surgery is a major risk factor for development of postoperative complications which effect both short and long-term outcome. Despite this 1 in 5 patients continue to smoke before their operation.

Project MURRAY is a trial comparing the effectiveness of personalised integrated smoking cessation delivered by trained health-care practitioners in the thoracic surgical pathway, and is a three part package of behaviour interventions and pharmacotherapy as per National Institute of Clinical Excellence (NICE)/ National Centre for Smoking Cessation Training (NCSCT) guidance which is supported by an adjunct web-based application. This is a pilot study to evaluate feasibility of a substantive trial and study processes in 5 adult thoracic centres including the trial coordinating site at the University Hospitals Birmingham NHS Foundation Trust. This is a multicentre feasibility study, with aim for equal weighting between the two arms of the integrated smoking cessation and an observation only group of usual care.

ELIGIBILITY:
Inclusion Criteria:

* Current tobacco smoker (smoked within the last 28 days)
* Major Thoracic Surgery (including both open and minimally invasive approach)
* Able to provide written informed consent
* At least 1 weeks' time to surgery
* Age over 18 years

Exclusion Criteria:

* Emergency thoracic surgery
* Inability to perform exhaled carbon monoxide (CO) measurements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-01-31 (Estimated); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment | 0 days from recruitment
  To establish the number of patients who agree to participate in the intervention as a proportion of those eligible to enter the study

SECONDARY OUTCOMES:
Integration of intervention | 0 days from recruitment, 1 day or surgery
  Integration of the intervention into the clinical pathway by time from decision to operate from study recruitment
Barriers to recruitment | 0 days from recruitment
  Descriptive reasons for non-participation from screening logs
Fine tune procedures and data capture forms | 0 days from recruitment, 1 day of surgery, 1 month after surgery
  To pilot data capture forms aiming for over 90% completion of important perioperative data for each patient
Smoking cessation in the intervention group | 1 day of surgery, 1 month after surgery
  To assess the proportion of patients who receive the intervention who have quit smoking
Smoking cessation in the usual care group | 1 day of surgery, 1 month after surgery
  To assess the proportion of patients in an observation only usual care group who have quit smoking
Variability of smoking cessation practices | 0 days from recruitment, 1 day of surgery, 1 month after surgery
  To define the variability of smoking cessation practices in all patients using the nicotine replacement usage questionnaire
Qualitative interview | 1 month after surgery
  To understand patients' experience of and engagement with the intervention, and any unintended consequences
  To establish whether the intervention is acceptable to thoracic surgery patients and staff, and investigate recommendations for optimisation in intervention delivery

CONTACTS AND LOCATIONS:
Overall Officials: Babu Naidu, MD, Principal Investigator — University of Birmingham

IPD SHARING:
Plan to Share IPD: Yes
Upon completion and publication of the study, individual participant data will be shared that underlie the results reported in study after de-identification. Additional related documents will be available including the study protocol, statistical analysis plan and an analytical code.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: This data will be available in the beginning 3 months and 5 years following article publication.
Access Criteria: To those who provide a methodologically sound proposal for analysis to achieve the aims in the approved proposal. All proposals should be directed to b.naidu@bham.ac.uk. To gain access requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Lugg ST, Kerr A, Kadiri S, Budacan AM, Farley A, Perski O, West R, Brown J, Thickett DR, Naidu B; Project MURRAY Investigators. Protocol for a feasibility study of smoking cessation in the surgical pathway before major lung surgery: Project MURRAY. BMJ Open. 2020 Nov 6;10(11):e036568. doi: 10.1136/bmjopen-2019-036568. PMID 33158819